CLINICAL TRIAL: NCT03701100
Title: The Effects of Bimodal Anodal Transcranial Direct Current Stimulation Over Bilateral Prefrontal Cortex on Illness Severity, Insight, Functional Outcomes, Quality of Life, Neurocognition and Heart Rate Variability (HRV) in Schizophrenia
Brief Title: The Effects of Bimodal tDCS on Illness Severity, Insight, Functional Outcomes, Neurocognition and HRV in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Hsin-An Chang, MD, Attending Psychiatrist, Department of Psychiatry, Principal Investigator, Assistant Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-103-03-002-3
Record Dates: First submitted 2018-10-06; First posted 2018-10-09 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia; Insight Impaired; Psychotic Symptoms; Schizoaffective Disorder; Neurocognitive Dysfunction; Autonomic Imbalance; Psychosocial Impairment; Quality of Life
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognition Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Direct current (DC) generated by a Eldith DC stimulator was bilaterally delivered through a pair of saline-soaked surface sponge electrodes (35 square centimeter). One anode was placed with the middle of the electrode over a point midway between International 10-20 electrode positions F3 and Fp1 (left dorsolateral prefrontal cortex and left prefrontal cortex). The other was located over a point midway between F4 and Fp2 (right dorsolateral prefrontal cortex and left prefrontal cortex). An extracephalic positions were used for the reference electrodes (cathodes) in order to avoid confounding effects from inhibitory cathodal effects at other cortical sites. The reference electrodes were placed on bilateral forearms. Stimulation was applied at an intensity of 2 milliampere (mA) (current density=1.14 A/square meter) for 20 min, twice-daily on 5 consecutive weekdays (total charge density=2736 C/square meter).
Who Masked: Participant, Outcomes Assessor
Masking Description: In sham stimulation, the current was turned on for 30 sec and then ramped down to 0 mA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Direct current (DC) generated by a Eldith DC stimulator was bilaterally delivered through a pair of saline-soaked surface sponge electrodes (35 square centimeter). One anode was placed with the middle of the electrode over a point midway between International 10-20 electrode positions F3 and Fp1 (left dorsolateral prefrontal cortex and left prefrontal cortex). The other was located over a point midway between F4 and Fp2 (right dorsolateral prefrontal cortex and left prefrontal cortex). The reference electrodes were placed on bilateral forearms. Stimulation was applied at an intensity of 2 mA for 20 min, twice-daily on 5 consecutive weekdays. All patients in the active tDCS group were maintained on their antipsychotic medications throughout the study period.
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): In sham stimulation, the current was turned on for 30 sec and then ramped down to 0 mA. All patients in the sham tDCS group were maintained on their antipsychotic medications throughout the study period.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — tDCS

SUMMARY:
The study aimed to investigate the effects of bimodal anodal transcranial direct current stimulation (tDCS) over bilateral dorsolateral prefrontal cortex (DLPFC) on psychopathological symptoms, insight, psychosocial functioning, neurocognitive function and heart rate variability (HRV) in schizophrenia patients

DETAILED DESCRIPTION:
Transcranial direct current stimulation encompasses the induction of a relatively weak constant current flow through the cerebral cortex via scalp electrodes . Dependent on stimulation polarity, this results in a modulation of cortical excitability and spontaneous neural activity.The technique was established in the 1950s and 1960s primarily in animals. In these early studies it was shown that subthreshold DC stimulation increases spontaneous neuronal activity if the anode is placed above or within the cortex, while exposure to cathodal polarity results in reduced activity. This is caused by a subthreshold membrane depolarization by anodal and a hyperpolarization by cathodal stimulation. It was demonstrated in humans that the after-effects of tDCS depend on modifications of N-methyl-D-aspartate (NMDA) receptor-efficacy. The after-effects of tDCS are blocked by the NMDA receptor antagonist dextromethorphan, and prolonged by the partial NMDA receptor-agonist D-cycloserine. This tDCS polarity-dependent alteration of NMDA receptor function seems to be initiated by the respective membrane potential shift and probably by the accompanying cortical activity modification,because it is prevented by the sodium channel blocker carbamazepine. Intraneuronal calcium concentration also contributes, because calcium channel antagonists eliminate the excitability-enhancing after-effects of anodal tDCS. Recently, unimodal anodal tDCS over left dorsolateral prefrontal cortex (DLPFC) has been found to improve psychopathological symptoms, cognitive deficits and insight of schizophrenia and also strengthen cardiac autonomic function in healthy subjects. Further studies using bimodal anodal tDCS over bilateral dorsolateral prefrontal cortex (DLPFC) and prefrontal cortex are needed.

Study design: randomized double-blind, sham-controlled study design.

Participants: 60 patients having a diagnosis of schizophrenia or schizoaffective were randomly allocated to receive 20 minutes of active 2-mA tDCS or sham stimulation twice a day on 5 consecutive weekdays. These participants were assessed at baseline, after intervention and in a three-months follow-up.

Active or sham stimulation: The present study used bimodal anodal tDCS over bilateral dorsolateral prefrontal cortex (DLPFC) and prefrontal cortex. One anode was placed with the middle of the electrode over a point midway between International 10-20 electrode positions F3 and Fp1 (left dorsolateral prefrontal cortex and left prefrontal cortex). The other was located over a point midway between F4 and Fp2 (right dorsolateral prefrontal cortex and left prefrontal cortex). An extracephalic positions were used for the reference electrodes (cathodes) in order to avoid confounding effects from inhibitory cathodal effects at other cortical sites. The reference electrodes were placed on bilateral forearms.

Others: see Arms and Interventions, Eligibility Criteria or Outcome Measures.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible participants aged 20-65 with DSM-IV-TR-defined schizophrenia or schizoaffective disorder.
2. Duration of illness ≧ 1 year.
3. Being on an adequate therapeutic dose of antipsychotics and clinically stable (nonacute phase of illness) but symptomatic for at least 4 weeks prior to enrolment as defined by Clinical Global Impression-Severity of Illness scale (CGI-S) score ≦ 4 (at both screening and baseline).
4. Agreement to participate in the study and provide the written informed consent.

Exclusion Criteria:

1. Having current psychiatric comorbidity or active substance use disorder, in exception to caffeine and/or tobacco.
2. Having history of seizures.
3. Having contraindications for tDCS, e.g., implanted brain medical devices or metal in the head.
4. Having history of intracranial neoplasms or surgery, or a history of severe head injuries or cerebrovascular diseases.
5. Pregnancy or breastfeeding at enrollment.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Changes from baseline scores of Positive and Negative Syndrome Scale (PANSS) at the timepoint immediately after tDCS, at one month and three months after tDCS. | Three months
  A clinician-administered rating scale to measure the severity of psychopathological symptoms of the patients with schizophrenia spectrum disorder. The patient is rated from 1 to 7 on 30 different symptom items. All items scores are summed up to yield a total PANSS score, which ranges from 30 to 210. A higher score indicates greater psychopathological symptom severity. Then, five main symptom dimension subscales of PANSS can be calculated from 26 of 30 items of PANSS: positive (5 items, score 5-35) , negative (8 items, score 8-56), grandiosity/excitement (4 items, score 4-28), disorganization (5 items, score 5-35), and depression (4 items, score 4-28).

SECONDARY OUTCOMES:
Changes from baseline scores at Personal and Social Performance scale (PSP) at the timepoint immediately after tDCS, at one month and three months after tDCS. | Three months
  A clinician-administered rating scale to measure the psychosocial functioning of the patients with schizophrenia spectrum disorder. The PSP scale measures psychosocial functioning within four domains: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior.The patient is rated from 1 to 6 on each item of the four domains. A higher score indicates greater psychosocial functioning in any of the four domains. The final global score is defined according to a summary instruction table. This scale provides a single, overall rating from 1 to 100, where a higher score represents better personal and social function.
Changes from baseline scores of the Global Assessment of Functioning (GAF) Scale of the DSM-IV at the timepoint immediately after tDCS, at one month and three months after tDCS. | Three months.
  GAF is a numeric scale used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of an individual, e.g., how well one is meeting various problems-in-living. Scores range from 100 (extremely high functioning) to 1 (severely impaired). GAF serves as a valid tool of assessing global psychosocial and occupational functioning for schizophrenia patients.
Changes from baseline scores of the Clinical Global Impression (CGI) rating scales at the timepoint immediately after tDCS, at one month and three months after tDCS. | Three months.
  Illness severity was assessed with the Clinical Global Impression (CGI) rating scales. The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. The patient is rated from 1 to 7 and a higher score indicates greater illness severity.
Changes from baseline scores of the self-reported version of the graphic personal and social performance scale (SRG-PSP) at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  The SRG-PSP is a self-rating scale of proven validity and reliability, comprising both male and female versions of cartoon-like pictures that are derived from the narrative text of the four domains of Personal and Social Performance (PSP) scale including the sub-items of socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behaviour.
Changes from baseline scores of the abbreviated version of the Scale to Assess Unawareness in Mental Disorder in schizophrenia (SUMD) at the timepoint immediately after tDCS, at one month and three months after tDCS. | Three months.
  An expert-rating scale based on a patient interview to measure patients' clinical insight. The abbreviated version of SUMD comprises 9 items measuring current states of awareness as follows: (1) a mental disorder, (2) consequences of a mental disorder, (3) effects of drugs, (4) hallucinatory experiences, (5) delusional ideas, (6) disorganized thoughts, (7) blunted affect, (8) anhedonia, and (9) lack of sociability. Scores on each item range from 0 to 3. A score of 0 indicates 'not applicable'; 1, 'aware'; 2, 'somewhat aware/unaware' and 3, 'severely unaware.' Based on the 3 dimensions approach of the abbreviated version of SUMD, the scores on the items 1-3, 4-6 and 7-9 were averaged to obtain the dimension score of 'awareness of the disease', 'awareness of positive symptoms', and 'awareness of negative symptoms', respectively. All dimension scores were linearized on a 0-100 scale, with 0 and 100 indicating the lowest and highest level of unawareness, respectively.
Changes from baseline scores of the Taiwanese version of the Beck Cognitive Insight Scale (BCIS) at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  Cognitive insight was measured by the Taiwanese version of the Beck Cognitive Insight Scale (BCIS), a self-reported instrument comprising 15 items.The Taiwanese BCIS is composed of 2 subscales including reflective attitude (9 items) and certain attitude (6 items). We obtained a R-C (reflective attitude minus certain attitude) index of the Taiwanese BCIS, representing the measurement of cognitive insight by subtracting the score of the certain attitude subscale from that of the reflective attitude subscale. Lower R-C index scores indicate poorer cognitive insight.
Changes from baseline scores of the Taiwanese version of the Self-Appraisal of Illness Questionnaire (SAIQ) at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  The Taiwanese version of the Self-Appraisal of Illness Questionnaire (SAIQ) was used to assess attitudes toward mental illness and experience of psychiatric treatment.This self-administered tool was composed of 17 items. The patients rated the extent to which they agreed with each statement of the item by using a four-point Likert scale, ranging from 1, ''do not agree at all'', to 4, ''completely agree''. Whether the scale score is in order from least to most or from the most to least depends on the content of the item statement. The total score of SAIQ ranges from 17 to 68. This translated SAIQ comprises a three-factor explanation. The three factors correspond to worry (score 7-28), the need for treatment (score 5-20), and presence/outcome (score 5-20) subscales. Higher SAIQ subscale scores indicate more awareness of mental illness.
Changes from baseline scores of the self-administered WHOQOL-BREF at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  The overall quality of life (QoL) and the specific domains of QoL was measured with the self-administered World Health Organization Questionnaire on Quality of Life: Short Form-Taiwan version (WHOQOL-BREF) which was developed by the WHO in 1998 and was adapted to Taiwan's culture. The WHOQOL-BREF is of well-established validity and reliability, containing 28 five-point Likert items that assessed general (two items) and four specific domains of QoL, including 7 items in physical health, 6 in psychological, 4 in social relationships, and 9 in environmental domains. Higher scores indicate a better QoL.
Changes from baseline results of Digit span (forward and backward) at the timepoint immediately after tDCS and at one month after tDCS. | One month
  A test to measure the capacity of working memory of the patients.
Changes from baseline results of Finger tapping test at the timepoint immediately after tDCS and at one month after tDCS. | One month
  A neuropsychological test that examines motor functioning, specifically, motor speed and lateralized coordination.
Changes from baseline results of Continuous Performance (CPT, version 2.0) at the timepoint immediately after tDCS and at one month after tDCS. | One month
  A neuropsychological test that examines the performance of prefrontal-mediated task.
Changes from baseline results of Wisconsin Card Sorting Test (WCST) at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  A neuropsychological test of "set-shifting", i.e. the ability to display flexibility in the face of changing schedules of reinforcement.
Changes from baseline results of Trail Making Test (TMT) at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  A neuropsychological test of visual attention and task switching.
Changes from baseline results of Tower of London test at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  A neuropsychological test for the assessment of executive functioning specifically to detect deficits in planning, which may occur due to a variety of medical and neuropsychiatric conditions.
Changes from baseline heart rate variability (HRV) at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  An index of autonomic functioning.
Changes from baseline scores of the Mini-Mental State Examination (MMSE) at the timepoint immediately after tDCS, at one month and three months after tDCS. | Three months.
  Global cognition was assessed with the Mini-Mental State Examination (MMSE).

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-An Chang, M.D., Principal Investigator — Tri-Service General Hospital, National Defense Medical Center
Locations (1):
- Tri-service general hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang CC, Kao YC, Chao CY, Tzeng NS, Chang HA. Examining bi-anodal transcranial direct current stimulation (tDCS) over bilateral dorsolateral prefrontal cortex coupled with bilateral extracephalic references as a treatment for negative symptoms in non-acute schizophrenia patients: A randomized, double-blind, sham-controlled trial. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Jan 10;96:109715. doi: 10.1016/j.pnpbp.2019.109715. Epub 2019 Jul 27. PMID 31362034